CLINICAL TRIAL: NCT05640804
Title: A Bioequivalence Study Between the Generic Dasatinib Tablet and Reference Product in Vivo
Brief Title: A Bioequivalence Study of Dasatinib Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZDTQ-BE-2017-DSTN
Record Dates: First submitted 2022-11-30; First posted 2022-12-07 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Myelogenous, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTTTQ Dasatinib tablet (Experimental): Subjects receive CTTQ dasatinib tablet under fasting/fed
  Interventions: Drug: CTTQ Dasatinib tablet
- Sprycel Sprycel (Experimental): Subjects receive Sprycel under fasting/fed
  Interventions: Drug: Sprycel Dasatinib tablet

INTERVENTIONS:
Drug: CTTQ Dasatinib tablet — Dasatinib tablet is an oral tyrosinekinase inhibitor produced by Chia Tai Tianqing Pharmaceutical Group.
  Arms: CTTTQ Dasatinib tablet
Drug: Sprycel Dasatinib tablet — Sprycel Dasatinib tablet is an oral tyrosinekinase inhibitor produced by Bristol Myers Squibb.
  Arms: Sprycel Sprycel

SUMMARY:
This is a clinical study to evaluate the bioequivalence of dasatinib tablet produced by Chia Tai Tianqing Pharmaceutical Group Co., Ltd. and Sprycel® produced by Bristol Myers Squibb after single dose in healthy subjects, so as to provide reference for clinical evaluation and clinical medication; to observe the safety of the dasatinib tablet and the reference drug Sprycel® in healthy subjects under fasting and fed states.

ELIGIBILITY:
Inclusion Criteria:

* Subjects signed the informed consent form before the trial and fully understood the trial content, process and possible adverse reactions;
* Subjects were able to complete the study according to the requirements of the trial protocol;
* Subjects have no disease history of heart, liver, kidney, digestive tract, nervous system, mental disorders and metabolic disorders;
* Healthy male and female subjects at age of 18-55;
* Male subjects weighted ≥ 50 kg, female subjects weighted ≥ 45kg, and the body mass index (BMI) was18 kg/m2 to 28 kg/m2 (including the cutoff value).
* Normal or not clinical significant abnormal vital signs, physical examination, laboratory examination, ECG and imaging examination have;
* The female blood pregnancy test was negative, and the subjects (including male subjects) had no pregnancy plan from 2 weeks before administration to at least 1 month after the last dose of the study drug and voluntarily took effective contraceptive measures.

Exclusion Criteria:

* Subjects with the following diseases or with clinically significant abnormalities in clinical laboratory examinations or other clinical findings of clinical significance (including but not limited to gastrointestinal, kidney, liver, neurological, blood, endocrine, tumor, lung, immune, psychiatric, cardiovascular and cerebrovascular diseases);
* Subjects with known allergies to dasatinib or its excipients;
* Subjects smoked at least 5 cigarettes per day 3 months before screening;
* Subjects with a history of drug or alcohol abuse;
* Subjects who donated blood within 3 months before screening;
* Subjects who took any drugs that could change liver enzyme activity 28 days before taking the study drug;
* Subjects who have taken any drugs, vitamin products or herbal medicines within 14 days before clinical trial;
* Subjects who smoked and drank alcohol during the trial, or performed strenuous exercise before the trial;
* Subjects have taken the study drug and participated in other drug clinical trials within 2 months before the clinical trial;
* Subjects with abnormal vital sign results;
* Subjects with abnormal clinical medical investigation;
* Subjects who had clinically significant ECG abnormalities;
* Subjects with abnormal chest X-rays;
* Subjects with the positive results of Hepatitis (including hepatitis B and C), AIDS, and syphilis;
* Female subjects who were lactating or serum-positive for pregnancy;
* Those who screen positive for drugs or have a history of drug abuse in the past five years or have used drugs in the three months prior to the trial;
* Subjects with acute illnesses that occurred during the screening period or prior to study drug administration;
* Acute disease occurs during pre-study screening stage or before study medication
* Subjects with a history of peptic ulcer or intracranial hemorrhage;
* Subjects had any disease that increased the risk of bleeding,
* Subjects were unable to comply with ward management regulations;
* Subjects cannot complete the trial for personal reasons;
* Subjects judged unsuitable for participating in this trial by other investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Maximum (peak) plasma drug concentration is a Pharmacokinetic parameter
Area under the plasma concentration-time curve from time zero to time t (AUC0-t) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Area under the plasma concentration-time curve from time zero to time t is a Pharmacokinetic parameter
The area under the plasma concentration curve from 0 to infinity (AUC0-∞) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  The area under the plasma concentration curve from 0 to infinity

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Time to reach maximum (peak) plasma concentration following drug administration
Elimination half-life (t1/2) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  The time required for the highest concentration of the drug in plasma to decrease by half
Apparent end elimination rate constant (λz) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Terminal disposition rate constant/terminal rate constant
Apparent volume of distribution (Vd/F) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Apparent volume of distribution after oral administration
Apparent total body clearance (CL/F) | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Apparent total clearance of the drug from plasma after oral administration
Relative bioavailability | 1 hour before administration and 15, 30, 45 minutes, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24 hours after administration.
  Bioavailability (systemic availability of the administered dose)
Adverse Event | Up to day 11
  Adverse events of subjects occured during the trial
Serious Adverse Event | Up to day 11
  Serious Adverse events of subjects occured during the trial
Body temperature | Up to day 11
  Monitor the body temperature of subjects and report abnormal body temperature
Pulse | Up to day 11
  Monitor the pulse of subjects and report abnormal pulse
Blood pressure | Up to day 11
  Monitor the blood pressure of subjects and report abnormal blood pressure
CTCAE v5.0 | Up to day 11
  The Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 (physical examination)
The Number of participants with abnormal laboratory examinations | Up to day 11
  laboratory examination, such as liver function, kidney function, coagulation function, blood routine, urine routine

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Changchun University of Traditional Chinese Medicine, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Xue J, Su Z, Cui Y, Liu G, Yang W, Liu Z, Chen J, Ren Q, Yu S, Cheng Y, Zhou Y, Wang W, Chen X, Qu D, Deng Q, Zhao Y, Yang H. Pharmacokinetics and safety of dasatinib and its generic: a phase I bioequivalence study in healthy Chinese subjects. Expert Opin Investig Drugs. 2023 Mar;32(3):263-270. doi: 10.1080/13543784.2023.2179481. Epub 2023 Feb 18. PMID 36757390